CLINICAL TRIAL: NCT02940418
Title: The Use of Mesenchymal Stromal Cells (MSC) in Type 1 Diabetes Mellitus in Adult Humans: Phase I Clinical Trial
Brief Title: Use of Stem Cells in Diabetes Mellitus Type 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sophia Al-Adwan (Other)
Responsible Party: Sponsor-Investigator, Sophia Al-Adwan, Biologist, PhD, University of Jordan
Organization: University of Jordan (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1DM.UJCTC
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Diabetes Mellitus; Type 1; Adipose derived mesenchymal stem cells
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose 1 mil/kg (Active Comparator): Adipose mesenchymal cells with bone marrow mononuclear cells.
  Two doses with a 6 month interval of allogenic Adipose mesenchymal cells +1 mil/kg of autologous bone marrow mononuclear cells will be injected intravenously.
  Interventions: Biological: Adipose mesenchymal cells with bone marrow mononuclear cells
- Dose 10 mil/kg (Active Comparator): Adipose mesenchymal cells with bone marrow mononuclear cells.
  Two doses with a 6 month interval of allogenic Adipose mesenchymal cells +10 mil/kg of autologous bone marrow mononuclear cells will be injected intravenously.
  Interventions: Biological: Adipose mesenchymal cells with bone marrow mononuclear cells

INTERVENTIONS:
Biological: Adipose mesenchymal cells with bone marrow mononuclear cells — Allogenic adipose-derived mesenchymal cells with autologous bone marrow mononuclear cells will be injected.

SUMMARY:
Allogenic adipose derived mesenchymal stem cells will be injected into patients newly diagnosed with type 1 Diabetes Mellitus

DETAILED DESCRIPTION:
Adipose derived mesenchymal stem cells (ASCs) are to be collected from blood group O donor, cells will be passaged to passage 5.

Before release the sample will be subject to our release criteria which include: testing for any bacterial or fungal growth as well as endotoxin and mycoplasma. All these tests must be negative. In addition the cell count and viability (must be more than 80%) are done before release. Surface markers documentation is done on the cells before release using flow cytometry.

The cells should be infused within 2 hours of release. The dose to is to be repeated after 6 months of a total of two doses in patients. Tests and follow up are to be one at week 12, 24 and 36 when the study is stopped.

These cells will be injected intravenously into patients newly diagnosed with type 1 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients with Type 1 Diabetes Mellitus.
2. Age from 18 years to 35 years either gender.
3. Duration of disease: not exceeding 3 years unless C-peptide is not less than 0.5 ng/ml
4. C-Peptide at inclusion base line should not be less than 0.5 ng/ml
5. No clinical evidence of renal, retinal, vascular or skin complications
6. Body Mass Index not exceeding 30
7. Any HbA1c
8. At least one positive antibody either anti-Glutamic Acid Decarboxylase-65 or Insulinoma-Associated-2 Autoantibodies (anti-1A2)
9. Informed Consent by patient

Exclusion Criteria:

1. Age less than 18 years and more than 35 years
2. Pregnancy
3. Married women or women expected to be married within the study period
4. History of allergy, Cancer, bronchial asthma, liver disease or hepatitis
5. Diabetic coma or pre-coma current or recent within the last 2 months
6. C-Peptide less than 0.5 ng/ml
7. Disease duration more than 3 yrs.
8. Complication mentioned in 5 above in inclusion
9. Non-consenting patient or withdrawal of consent.
10. Bleeding disorders

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-19 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Safety of using allogenic ASC assessed by any adverse events | 6 months
  Patients will be assessed for any adverse events as a result of the injection.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Awidi, MD, Study Director — Cell Therapy Center
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided